CLINICAL TRIAL: NCT07324629
Title: A Phase II Clinical Study of Sacituzumab Tirumotecan in Participants With Locally Advanced or Metastatic Thymic Carcinoma With Treatment Failure After Platinum-Based Therapy
Brief Title: Sacituzumab Tirumotecan in Participants With Locally Advanced or Metastatic Thymic Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan Kelun-Biotech Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sichuan Kelun Pharmaceutical Research Institute Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SKB264-II-17
Record Dates: First submitted 2025-12-11; First posted 2026-01-07 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Thymic Carcinoma
MeSH Terms: conditions — Thymoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sac-TMT 5mg/kg Q2W (Experimental)
  Interventions: Drug: Sacituzumab tirumotecan

INTERVENTIONS:
Drug: Sacituzumab tirumotecan — Sacituzumab tirumotecan (Sac-TMT; also known as SKB264) for injection.

SUMMARY:
The goal of this clinical trial is to learn if drug Sac-TMT works to treat Thymic Carcinoma. It will also learn about the safety of Sac-TMT. The main questions it aims to answer are:

* How effective is drug Sac-TMT in treating Thymic Carcinoma?
* What adverse events (AEs) do participants have when taking drug Sac-TMT?

Participants will:

* Progress after at least one platinum-based chemotherapy treatment.
* Take drug Sac-TMT every 2 weeks.
* Take tumor response assessments every 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged ≥ 18 to ≤ 75 years at the time of signing the Informed Consent Form;
* Participants with histologically or cytologically confirmed thymic carcinoma, and locally advanced or metastatic thymic carcinoma who are not suitable for curative intent therapy;
* Participants with advanced thymic carcinoma who have progressed after at least one prior platinum-based chemotherapy;
* Able to provide a tumor tissue sample at the time of or after the diagnosis of locally advanced or metastatic tumor;
* At least one measurable target lesion that has not received radiotherapy according to RECIST v1.1;
* ECOG performance status score of 0 or 1;
* Expected survival ≥ 12 weeks;
* Adequate organ and bone marrow function.

Exclusion Criteria:

* Participants with histologically or cytologically confirmed thymoma or thymic neuroendocrine tumor;
* Participants with known metastases to meninges, brainstem metastases, spinal cord metastases and/or compression, active or untreated brain metastases;
* Participants with other malignant tumors within 3 years prior to the first dose;
* Presence of any of conditions or risk factors related to cardiovascular and cerebrovascular diseases;
* Uncontrolled systemic disease as judged by the investigator;
* History of interstitial lung disease/noninfectious pneumonitis requiring steroid therapy;
* Clinically severe pulmonary impairment due to lung disorder;
* Presence of active hepatitis B or hepatitis C;
* Known active tuberculosis;
* Known hypersensitivity to the study drug or any of its components.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-04 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
ORR | From enrollment to the end of treatment at 24 months
  To evaluate the objective response rate (ORR) of sac-TMT as assessed by the investigator based on RECIST v1.1.

SECONDARY OUTCOMES:
PFS | From enrollment to the end of treatment at 24 months
  To evaluate the progression-free survival (PFS) as assessed by the investigator based on RECIST v1.1.
OS | From enrollment to the end of treatment at 24 months
  To evaluate the overall survival (OS) of sac-TMT in participants with locally advanced or metastatic thymic carcinoma with treatment failure after platinum-based therapy.
Incidence and severity of AEs and SAEs, and abnormal laboratory values. | From enrollment to the end of treatment at 24 months
  To evaluate the safety of sac-TMT in participants with locally advanced or metastatic thymic carcinoma.
DCR | From enrollment to the end of treatment at 24months
  Duration of response (DOR) as assessed by the investigator based on RECIST v1.1.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, China